CLINICAL TRIAL: NCT00023907
Title: A Phase II Evaluation of Weekly Paclitaxel in the Treatment of Recurrent or Persistent Platinum and Paclitaxel-Resistant Ovarian or Primary Peritoneal Cancer
Brief Title: Paclitaxel in Treating Patients With Ovarian Epithelial Cancer or Primary Peritoneal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068875; GOG-0126N
Record Dates: First submitted 2001-09-13; First posted 2003-07-09 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2004-05

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Paclitaxel

INTERVENTIONS:
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of paclitaxel in treating patients who have recurrent or persistent ovarian epithelial cancer or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of paclitaxel in patients with recurrent or persistent platinum- and paclitaxel-resistant ovarian epithelial or primary peritoneal cancer.
* Determine the nature and degree of toxicity of this drug in these patients.

OUTLINE: Patients receive paclitaxel IV over 1 hour once weekly for 4 weeks. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 19-51 patients will be accrued for this study within 6-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed recurrent or persistent ovarian epithelial or primary peritoneal cancer
* Measurable disease

  * At least 1 lesion measured in at least 1 dimension

    * At least 20 mm by conventional techniques OR
    * At least 10 mm by spiral CT scan
* At least 1 target lesion

  * Tumors within a previously irradiated field considered non-target lesions
* Paclitaxel resistant

  * Treatment-free interval of less than 6 months duration after treatment with prior paclitaxel OR
  * Progression during prior paclitaxel-based therapy
* Platinum resistant or refractory

  * Treatment-free interval of less than 6 months duration after treatment with prior platinum OR
  * Progression during prior platinum-based therapy
* Ineligible for higher priority GOG protocol (any active GOG phase III protocol for the same patient population)

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* GOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection requiring antibiotics
* No other prior invasive malignancy within the past 5 years except nonmelanoma skin cancer
* No grade 2 or greater neuropathy (sensory and motor)

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 3 weeks since prior biologic or immunologic agents for cancer

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy for cancer and recovered
* Received at least 1 but no more than 2 prior platinum-based chemotherapy regimens containing carboplatin, cisplatin, or other organoplatinum compound for primary or recurrent disease
* Initial treatment may include high-dose therapy, consolidation, or extended therapy
* Received at least 1 prior paclitaxel-based chemotherapy regimen
* No prior paclitaxel or docetaxel with a schedule of less than a 3-week interval between doses
* No additional prior cytotoxic chemotherapy for recurrent or persistent disease, including retreatment with initial chemotherapy regimens

Endocrine therapy:

* At least 1 week since prior hormonal therapy for cancer
* Concurrent hormone replacement therapy allowed

Radiotherapy:

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy for cancer and recovered
* No prior radiotherapy to site(s) of measurable disease
* No prior radiotherapy to more than 25% of marrow-bearing areas

Surgery:

* At least 3 weeks since prior surgery for cancer and recovered

Other:

* At least 3 weeks since other prior therapy for cancer
* No prior anticancer treatment that would preclude study
* No concurrent amifostine or other protective reagents

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-07; Primary Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurie Markman, MD, Study Chair — The Cleveland Clinic
Locations (44):
- United States (44):
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Women's Cancer Center at Community Hospital of Los Gatos, Los Gatos, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Cancer Center, Orange, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Keesler Medical Center - Keesler Air Force Base, Keesler Air Force Base, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Southeast Gynecologic Oncology Associates, Knoxville, Tennessee
  - Genecologic Oncology Network, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin

REFERENCES:
- [Result] Gynecologic Oncology Group; Markman M, Blessing J, Rubin SC, Connor J, Hanjani P, Waggoner S. Phase II trial of weekly paclitaxel (80 mg/m2) in platinum and paclitaxel-resistant ovarian and primary peritoneal cancers: a Gynecologic Oncology Group study. Gynecol Oncol. 2006 Jun;101(3):436-40. doi: 10.1016/j.ygyno.2005.10.036. Epub 2005 Dec 2. PMID 16325893